CLINICAL TRIAL: NCT06517875
Title: A Phase 2 Open-label Study to Evaluate Momelotinib in Combination With Luspatercept in Participants With Transfusion Dependent Primary or Secondary Myelofibrosis
Brief Title: Study of Momelotinib in Combination With Luspatercept in Participants With Transfusion Dependent Myelofibrosis
Acronym: ODYSSEY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 220752; 2024-518225-15 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Primary Myelofibrosis; Myelofibrosis; Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: Momelotinib; Luspatercept; Primary Myelofibrosis; Secondary Myelofibrosis; JAK inhibitor; anemia transfusion; Ojjara; Omjjara; Reblozyl
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide; luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Momelotinib + Luspatercept (Experimental): Participants with transfusion dependent primary myelofibrosis or post- PV/ ET myelofibrosis that is JAKi naïve or JAKi experienced will receive momelotinib and luspatercept.
  Interventions: Drug: Momelotinib; Drug: Luspatercept

INTERVENTIONS:
Drug: Momelotinib — Momelotinib will be administered orally.
  Other Names: Ojjaara; CYT387
Drug: Luspatercept — Luspatercept will be administered subcutaneously.
  Other Names: REBLOZYL; ACE-536

SUMMARY:
The purpose of this Phase 2 study is to evaluate the efficacy and safety of momelotinib (MMB) in combination with luspatercept (LUSPA) in participants with transfusion dependence (TD) primary myelofibrosis (PMF) or Post-polycythemia vera (PV)/ essential thrombocythemia (ET) myelofibrosis (MF) who are either janus kinase (JAK) inhibitor (JAKi) naïve or experienced.

ELIGIBILITY:
Inclusion Criteria:

1. Is age ≥18 years.
2. Confirmed diagnosis of PMF in accordance with the World Health Organization (WHO) 2016 criteria, or Post-PV/ET myelofibrosis in accordance with the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria.
3. JAKi naïve or previously treated with either ruxolitinib or fedratinib for PMF or Post-PV/ET myelofibrosis for ≥90 days, or ≥28 days if JAKi therapy is complicated by RBC transfusion requirement of ≥4 units in 8 weeks, or Grade 3/4 AEs of thrombocytopenia, anemia, or hematoma.
4. High risk, intermediate-2, or intermediate-1 risk as defined by Dynamic International Prognostic Scoring System (DIPSS) [Passamonti, 2010] or DIPSS-plus [Gangat, 2011].
5. TD defined as requiring RBC transfusion ≥4 units or HgB < 8 g/dL in the 8 weeks prior to the first dose of study treatment. Only transfusions given when Hgb levels are ≤9.5 g/dL are counted towards TD. RBC transfusions given for clinically overt bleeding, or accident/injury (as assessed by the investigator) are not counted towards TD.

Exclusion Criteria:

1. History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (e.g., uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study intervention or result in inability to swallow oral medications.
2. Participants with an invasive malignancy or history of invasive malignancy other than the disease under study within the last 5 years.
3. Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, gastrointestinal bleeding, or thalassemia.
4. Uncontrolled intercurrent illness:

   1. Active uncontrolled infection (participants receiving outpatient antibacterial and/or antiviral treatments for infection that is under control or as infection prophylaxis may be included in the trial);
   2. Uncontrolled acute and chronic liver disease (e.g., Child-Pugh score ≥10) OR has current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. NOTE: Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) is acceptable if participant otherwise meets entry criteria.
5. Uncontrolled hypertension, defined as repeated elevations of systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, that is not resolved at the time of the first dose of study treatment.
6. Any of the following in conditions within 6 months prior to the first dose of study intervention:

   1. Unstable angina pectoris; OR
   2. Symptomatic congestive heart failure; OR
   3. Uncontrolled cardiac arrhythmia
7. QTc interval >450 msec or QTc >480 msec for participants with bundle branch block.
8. Participants with stroke, deep venous thrombosis, pulmonary or arterial embolism within 6 months prior to the first dose of study intervention.
9. History of porphyria.
10. Presence of peripheral neuropathy ≥Grade 2 per CTCAE v5.0.
11. Use of the following treatments within the time periods noted NOTE: All active anti-MF therapy must discontinue at least 1 week prior to the start of baseline MFSAF recording (Study Day -7):

    1. Active anti-MF therapy within 28 days or 5 half-lives, whichever is shorter (exception is prior JAKi therapy).
    2. Steroid use for the treatment of myelofibrosis is prohibited within 14 days prior to the first dose of study treatment until discontinuation of study treatment. Supportive care including steroids for non-myelofibrosis indications may be used.
    3. Potent cytochrome P450 3A4 (CYP3A4) inducers, except for rifampin and rifampicin, within 14 days prior to the first dose of study intervention.
    4. Any prior investigational agent for myelofibrosis within 4 weeks prior to the first dose of study treatment.
    5. Erythropoiesis stimulating agent (ESA) within 4 weeks prior to the first dose of study treatment.
    6. Splenic irradiation within 3 months prior to the first dose of study treatment.
12. Prior treatment with MMB.
13. Prior treatment with luspatercept or sotatercept.
14. Prior splenectomy.
15. Inability or unwillingness to comply with the protocol restrictions on myelofibrosis therapy and other medications prior to and during study treatment.
16. Unresolved non-hematologic toxicities from prior therapies that are >Grade 1 per CTCAE v5.0 unless otherwise specified.
17. Known positive status for human immunodeficiency virus (HIV).
18. Hepatitis A, B, or C status as defined below:

    1. Chronic active or acute viral hepatitis A.
    2. Active Hepatitis B infection indicated by the presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to the first dose of study intervention.
    3. Positive hepatitis C antibody test result at screening or within 3 months before the first dose of study intervention. NOTE: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative hepatitis C ribonucleic acid (RNA) test is obtained.
19. Women who are already pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with TI Response by Week 24 | Up to Week 24
  TI response is defined as not requiring red blood cell (RBC) transfusion (except in the case of clinically overt bleeding) for any ≥12-week interval.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation | Up to approximately 36 weeks
Number of Participants with Clinically Important Changes in Laboratory Parameters, Vital Signs, and Eastern Cooperative Oncology Group (ECOG) Performance Status | Up to Week 24
Percentage of Participants with TI at the End of Week 24 | Up to Week 24
  TI was defined as not requiring RBC transfusion (except in the case of clinically overt bleeding) for ≥12 weeks preceding Week 24, with all hemoglobin (Hgb) levels during the ≥12-week interval of ≥8 g/dL (except in the case of clinically overt bleeding).
Plasma Concentration of MMB | Up to Week 24
Plasma Concentration of Morpholino Lactam (M21) | Up to Week 24

CONTACTS AND LOCATIONS:
Locations (14):
- GSK Investigational Site, Nashville, Tennessee, United States
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (7):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poitiers
- Italy (2):
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Roma
- Spain (2):
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: No